CLINICAL TRIAL: NCT06118619
Title: A Multicenter Clinical Trial of Recombinant Human Interferon Gamma (Ingaron) in Pulmonary Tuberculosis
Brief Title: A Multicenter Clinical Trial of Ingaron in Pulmonary Tuberculosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SPP Pharmaclon Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: GAM2022
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Respiratory Tuberculosis
Keywords: Respiratory tuberculosis; interferon gamma
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Interferon-gamma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Ingaron 500,000 IU intramuscularly 1 time per day daily or every other day for 2 months (60 days) - a total of 30 or 60 injections + basic anti-tuberculosis therapy
  Interventions: Drug: Interferon-Gamma
- No Intervention: only basic anti-tuberculosis therapy

INTERVENTIONS:
Drug: Interferon-Gamma — received by microbiological synthesis; specific antiviral activity on cells is 2x10*7 Units per mg of protein
  Other Names: Ingaron; Interferon gamma human recombinant
  Groups: Experimental

SUMMARY:
The main purpose of testing: To confirm the effectiveness and safety of the drug Ingaron when used in patients hospitalized at the research center for various reasons.

DETAILED DESCRIPTION:
Monitoring of a patient in a hospital is carried out daily by the attending physician during the entire period of the patient's stay at the research center. When prescribing the drug Ingaron, the researcher must follow the instructions for use of the drug. As part of 4 control observations to assess effectiveness and safety:

* 1st on the 1st day of using the drug Ingaron and starting anti-tuberculosis therapy
* 2nd on the 30th - 31st day of therapy
* 3rd after 2 months of therapy
* 4th (final) after 3 months of follow-up After each of the 3 visits, the research doctor saves the data necessary for further evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 78 years inclusive
2. Bacterioscopically and/or molecularly genetically verified diagnosis of tuberculosis
3. Stay in the intensive phase of treatment
4. Consent to inpatient anti-tuberculosis therapy until the end of participation in clinical observation

Exclusion Criteria:

1. Serious condition
2. Pregnancy
3. Breastfeeding
4. Treatment with immunomodulatory drugs before inclusion in the observation program
5. Presence of medical history of an allergic reaction or individual intolerance to the drug Ingaron
6. Severe diseases of the liver, kidneys (creatinine more than 150 mmol/l)
7. Presence of contraindications to the administration of the drug Ingaron
8. Patients with HIV infection with a CD4 lymphocyte count less than 350 cells/ml

Ages: 18 Years to 78 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of abacillated patients | 1 month
  Proportion of abacillated patients according to fluorescence microscopy
Proportion of abacillated patients | 1 month
  Proportion of abacillated patients according to culture data
Proportion of abacillated patients | 2 month
  Proportion of abacillated patients according to fluorescence microscopy
Proportion of abacillated patients | 2 month
  Proportion of abacillated patients according to culture data

SECONDARY OUTCOMES:
Proportion of patients who died | 5 month
  deaths associated with HIV infection and/or tuberculosis
Proportion of patients who required a change in therapy | 5 month
  Proportion of patients who required a change in therapy due to ineffectiveness
Proportion of patients with adverse reactions | 5 month
  Proportion of patients with adverse reactions, including those who required changes in therapy due to intolerance
Changes in the level of CD4 lymphocytes and HIV viral load in the blood | 5 month
  Changes in the level of CD4 lymphocytes and HIV viral load in the blood (Proportion of patients with a CD4 level less than 350 cells/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly I Saulin, Master, Study Director — SPP Pharmaclon Ltd.
Locations (13):
- Russia (13):
  - Astrakhan Oblast Tuberculosis Clinic, Astrakhan, Astrakhan Oblast
  - Tuberculosis Clinic of the Republic of Bashkortostan, Ufa, Bashkortostan Republic
  - Tuberculosis Clinic of the Chuvash Republic, Cheboksary, Chuvashskaya Respublika
  - Leningrad Oblast Tuberculosis Clinic, Slantsy, Leningradskaya Oblast'
  - Leningrad Oblast Tuberculosis Hospital in Tikhvin, Tikhvin, Leningradskaya Oblast'
  - Clinical Phthisiopulmonological Medical Center, Perm, Perm Krai
  - Ryazan Oblast Tuberculosis Clinic, Ryazan, Ryazan Oblast
  - Sverdlovsk Oblast Clinical Medical Center of Phthisiopulmonology and Infectious Diseases, Yekaterinburg, Sverdlovsk Oblast
  - Republican Tuberculosis Clinic, Kazan', Tatarstan Republic
  - Volgograd Oblast Tuberculosis Clinic, Volgograd, Volgograd Oblast
  - N. S. Pokhvisneva Voronezh Oblast Clinical Tuberculosis Dispensary, Voronezh, Voronezh Oblast
  - Yaroslavl regional tuberculosis clinic, Yaroslavl, Yaroslavl Oblast
  - City tuberculosis clinic, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Izosimova VE, Barmina NA, Zharikova MP, Alekseyev OY, Ryzhkova OA, Sayfulin MH, Popova NA, Andreyev MA, Gagarina SG, Rysdauletova RM, Kamaeva NG, Samoylova AG, Romanova MI. A Clinical Multicenter Trial of Recombinant Human Interferon Gamma in Tuberculosis (GAM2022): Experience with the Use of Human Recombinant Interferon Gamma in TB Practice. Infect Disord Drug Targets. 2025;25(6):e18715265329137. doi: 10.2174/0118715265329137250102103507. PMID 39871554